CLINICAL TRIAL: NCT06896071
Title: Project SOLVE and Rangatahi in Aotearoa: Evaluating a Digital Single-Session Intervention for Adolescent Mental Health in New Zealand Through a School-based Randomised Controlled Trial
Brief Title: Evaluating a Digital Single-session Intervention for Adolescent Mental Health in New Zealand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Waikato (Other)
Collaborators: Whau Mental Health Foundation (New Zealand) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HREC(Health)2024#60
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Project SOLVE (Experimental): In this arm, participants will complete Project SOLVE.
  Interventions: Behavioral: Project SOLVE
- Project Success (Active Comparator): In this arm, participants will complete Project Success.
  Interventions: Behavioral: Project Success

INTERVENTIONS:
Behavioral: Project SOLVE — Project SOLVE is a 30-minute self-guided online activity that includes an introduction to problem solving and which types of problems might be most appropriate for this skill; a description of how the brain facilitates problem solving; vignettes demonstrating how older adolescents have solved their problems; scientific evidence that problem solving can work; practice exercises; and activities to encourage the use of problem solving in daily life. The intervention teaches students how to solve problems via the "SOLVE" framework (i.e., Saying what the problem is; One goal to aim for; Listing some solutions; Voting for the best solution; Exploring what works).
  Arms: Project SOLVE
Behavioral: Project Success — Project Success is comparable to Project SOLVE in format and length (i.e., a 30 minute online, self-guided intervention) and teaches young people three strategies to reach their academic goals: how to take effective notes, how to break big assignments down into smaller tasks, and how to ask trusted others for help.
  Arms: Project Success

SUMMARY:
Currently, one in five rangatahi (young people) in Aotearoa report difficulty accessing support for their mental health concerns. This treatment gap has prompted academics and clinicians to consider whether online and/or school-based interventions can increase access to evidence-based mental health care.

This research is a randomised controlled trial to evaluate the effectiveness of Project SOLVE, an online problem-solving intervention, compared to Project Success, an activity that teaches young people study skills. Underdeveloped problem-solving skills have been associated with varying presentations of mental distress, including depression, hopelessness, and suicidal ideation. This association has meant problem solving is often featured as a core component of therapeutic interventions, and strengthening problem solving skills has been shown to improve clinical outcomes in youth who experience mental health concerns.

For these reasons, the investigators hope that Project SOLVE will support the development of problem solving in rangatahi in Aotearoa and have a positive effect on their proximal and longitudinal mental health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any Year 9 student (ages 12-14 years old) at a participating school who provides assent.

Exclusion Criteria:

* Any Year 9 student (ages 12-14 years old) at a participating school who does not provide assent and/or whose parent/caregiver does not provided consent.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Internalising and externalising symptoms | Immediately pre-intervention, immediately post-intervention and 12 weeks post-intervention
  Internalising and externalising symptoms will be measured using the Behaviour and Feelings Survey.

SECONDARY OUTCOMES:
Social Problem Solving Skills | Immediately pre-intervention and 12 weeks post-intervention
  Social problem solving will be measured by the Social Problem-Solving Inventory - Revised Short-Form.
General Self-Efficacy | Immediately pre-intervention, immediately post-intervention and 12 weeks post-intervention
  Self-efficacy will be measured using the General Self-Efficacy Scale.
Hope | Immediately pre-intervention, immediately post-intervention and 12 weeks post-intervention
  Hope will be measured using the Child Hope Scale.
Hopelessness | Immediately pre-intervention, immediately post-intervention and 12 weeks post-intervention
  Hopelessness will be measured using the Beck Hopelessness Scale - Shortened.
Well-Being | Immediately pre-intervention and 12 weeks post-intervention
  Well-being will be measured using the World Health Organisation Well-Being Index.
Educational Self-Efficacy | Immediately pre-intervention, immediately post-intervention and 12 weeks post-intervention
  Educational self-efficacy will be measured using the Educational Self-Efficacy Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan T Blind, BA(Hon), Principal Investigator — University of Waikato
Locations (1):
- St Peter's School Cambridge, Cambridge, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fenwick-Smith A, Dahlberg EE, Thompson SC. Systematic review of resilience-enhancing, universal, primary school-based mental health promotion programs. BMC Psychol. 2018 Jul 5;6(1):30. doi: 10.1186/s40359-018-0242-3. PMID 29976252
- [Background] Thabrew H, Stasiak K, Hetrick SE, Wong S, Huss JH, Merry SN. E-Health interventions for anxiety and depression in children and adolescents with long-term physical conditions. Cochrane Database Syst Rev. 2018 Aug 15;8(8):CD012489. doi: 10.1002/14651858.CD012489.pub2. PMID 30110718
- [Background] Ludin N, Holt-Quick C, Hopkins S, Stasiak K, Hetrick S, Warren J, Cargo T. A Chatbot to Support Young People During the COVID-19 Pandemic in New Zealand: Evaluation of the Real-World Rollout of an Open Trial. J Med Internet Res. 2022 Nov 4;24(11):e38743. doi: 10.2196/38743. PMID 36219754
- [Background] Sutcliffe K, Ball J, Clark TC, Archer D, Peiris-John R, Crengle S, Fleming TT. Rapid and unequal decline in adolescent mental health and well-being 2012-2019: Findings from New Zealand cross-sectional surveys. Aust N Z J Psychiatry. 2023 Feb;57(2):264-282. doi: 10.1177/00048674221138503. Epub 2022 Dec 1. PMID 36453262
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Background] Schleider JL, Mullarkey MC, Fox KR, Dobias ML, Shroff A, Hart EA, Roulston CA. A randomized trial of online single-session interventions for adolescent depression during COVID-19. Nat Hum Behav. 2022 Feb;6(2):258-268. doi: 10.1038/s41562-021-01235-0. Epub 2021 Dec 9. PMID 34887544